CLINICAL TRIAL: NCT00834314
Title: Vacuum-Therapy in Open Abdomen Treatment - Randomized Pilot-trial Comparing Fascial Closure and Survival With "Vacuum-Pack"-Technique vs. "Abdominal Dressing"
Brief Title: Randomized Pilot Study Comparing Two Vacuum-wound-dressings for Open Abdomen Treatment
Acronym: ABDOVAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: extended obligations of amended medical device law in Germany 2010 did not allow to continue and complete the trial due to budget limitation
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Prof Dr. Stefan Post, Prof. Dr., Director of Surgical Department, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-291 M-MA
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Open Abdomen; Temporary Abdominal Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vacuum-pack (Experimental): see Interventions
  Interventions: Procedure: Vacuum-Pack-technique for temporary abdominal closure
- Abdominal dressing (Active Comparator): see Interventions
  Interventions: Procedure: Abdominal-dressing-technique for temporary abdominal closure

INTERVENTIONS:
Procedure: Vacuum-Pack-technique for temporary abdominal closure — Negative-pressure-wound-therapy applying a method described by Brock, Barker et al 1995: "Temporary Closure of Open Abdominal Wounds - the Vacuum Pack" (see citations).
  Arms: Vacuum-pack
Procedure: Abdominal-dressing-technique for temporary abdominal closure — Negative-pressure-wound-therapy for temporary abdominal closure applying a device of KCI International (V.A.C.® Abdominal Dressing System). see: http://www.kci-medical.com/kci/corporate/kcitherapies/vactherapy/dressings/abdominal/#
  Other Names: V.A.C.® Abdominal Dressing System
  Arms: Abdominal dressing

SUMMARY:
The primary purpose of the study is to determine whether two vacuum-wound-dressing techniques (the so called "abdominal dressing" versus "vacuum-pack-technique") are equally effective in the treatment of open abdomen.

Secondary purpose is the comparison of feasibility and economic aspects.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for open-abdomen-treatment by responsible consultant surgeon where vacuum-technique is judged technically possible

Exclusion Criteria:

* Technical reasons
* unjustified risk-benefit-ratio of manipulations necessary for application of vacuum-pack-technique or abdominal-dressing-technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Failure of delayed abdominal fascial closure (non-prevented ventral hernia) and/or in-hospital-death of any cause (combined primary outcome) | until end of vacuum-therapy or death

SECONDARY OUTCOMES:
vacuum-therapy-related morbidity/complications | until hospital dismissal or death
length of vacuum-therapy | until end of vacuum-therapy or death
costs of vacuum-therapy | until end of vacuum-therapy or death
total length of ICU-stay | until end of ICU-therapy or death
post-dismissal health-related quality of life (SF36 and EQ-5D questionnaire) | 12 weeks after hospital dismissal
recurrent hernia/abdominal wall dehiscence after initial facial closure during hospital stay | 12 weeks post hospital dismissal

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Post, Prof. Dr., Principal Investigator — University Medical Center Mannheim, Germany, Surgical Department
Locations (1):
- University Medical Centre - Surgical Department, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Brock WB, Barker DE, Burns RP. Temporary closure of open abdominal wounds: the vacuum pack. Am Surg. 1995 Jan;61(1):30-5. PMID 7832378
- [Background] Barker DE, Green JM, Maxwell RA, Smith PW, Mejia VA, Dart BW, Cofer JB, Roe SM, Burns RP. Experience with vacuum-pack temporary abdominal wound closure in 258 trauma and general and vascular surgical patients. J Am Coll Surg. 2007 May;204(5):784-92; discussion 792-3. doi: 10.1016/j.jamcollsurg.2006.12.039. Epub 2007 Mar 26. PMID 17481484
- See also: Description of abdominal-dressing-technique; KCI-International company — http://www.kci1.com/cs/Satellite?c=KCI_Product_C&childpagename=KCI1%2FKCILayout&cid=1229624985184&p=1229538260417&packedargs=locale%3Den_US&pagename=KCI1Wrapper